CLINICAL TRIAL: NCT03084237
Title: Double-blind, Randomized, Multicenter, Phase III Clinical Study to Compare the Efficacy and to Evaluate the Safety and Immunogenicity of Trastuzumab Biosimilar HLX02 and EU-sourced Herceptin® in Previously Untreated HER2 Overexpressing Metastatic Breast Cancer
Brief Title: Compare Efficacy, Safety and Immunogenicity of HLX02 and Herceptin in Previously Untreated HER2 +Overexpressing Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX02-BC01; 2016-000206-10 (EudraCT Number)
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX02+Docetaxel (Experimental): HLX02+Docetaxel
  Interventions: Biological: HLX02; Drug: docetaxel
- Herceptin®+Docetaxel (Active Comparator): Herceptin®+Docetaxel
  Interventions: Biological: Herceptin®; Drug: docetaxel

INTERVENTIONS:
Biological: HLX02 — 8 mg/kg administered intravenously over 90 minutes as a loading dose on Day 1, Cycle 1 then 6 mg/kg every 3 weeks for subsequent cycles.
  Arms: HLX02+Docetaxel
Biological: Herceptin® — 8 mg/kg administered intravenously over 90 minutes as a loading dose on Day 1, Cycle 1 then 6 mg/kg every 3 weeks for subsequent cycles
  Arms: Herceptin®+Docetaxel
Drug: docetaxel — 75 mg/m2 will be administered on Day 2, Cycle 1.then be given every 3 weeks on Day 1 of each subsequent cycle

SUMMARY:
This is a Phase III, double-blind, randomized multicenter study to compare the efficacy and to evaluate the safety and immunogenicity of HLX02 and European Union (EU)-sourced Herceptin® in patients with human epidermal growth factor receptor 2 (HER2)-positive, locally recurrent or previously untreated metastatic breast cancer.

DETAILED DESCRIPTION:
This is a Phase III, double-blind, randomized multicenter study to compare the efficacy and to evaluate the safety and immunogenicity of HLX02 and European Union (EU)-sourced Herceptin® in patients with human epidermal growth factor receptor 2 (HER2)-positive, recurrent or previously untreated metastatic breast cancer. Eligible patients will be assessed centrally for HER2 status and the presence of at least one measurable target lesion before randomization. Patients will undergo a tumor assessment for evaluation of response according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) every 6 weeks up to 24 weeks (regardless of the number of cycles actually given); thereafter, assessments will be done every 9 weeks (after Cycles 11, 14, and 17) or earlier in the case of clinical signs of progression.

ELIGIBILITY:
Inclusion Criteria

* Patients have voluntarily agreed to participate and given written informed consent.
* Male or female ≥18 years of age on day of signing the informed consent form (ICF).
* Histologically or cytologically confirmed adenocarcinoma of the breast.
* Recurrent disease not amenable to curative surgery or radiation therapy, or metastatic disease with an indication for a taxane-containing therapy.
* Availability of formalin-fixed paraffin-embedded (FFPE) tissue block from the primary tumor, or a metastatic lesion, to confirm HER2-positivity by the central laboratory, based on FISH amplification ratio ≥2.0 or IHC score 3+, and for hormone status (ER/PgR) determination (local or central laboratory). If not possible, a fresh biopsy is required.
* No prior systemic anticancer agent such as chemotherapy, biological or targeted agent for metastatic disease with the exception of hormonal therapy, which must be stopped at least 2 weeks before randomization. Use of herbal remedies or traditional Chinese medicines for anticancer, hematologic or liver function, or anti-infective treatment must be stopped at the time of the ICF signature (at least 2 weeks before randomization).
* For patients with recurrent disease, prior neo-/adjuvant therapy containing trastuzumab and/or lapatinib must have been stopped at least 12 months before the diagnosis of recurrent (local or metastatic) disease. If trastuzumab/lapatinib was not used, prior neo-/adjuvant therapy with a taxane must have been stopped at least 6 months before the diagnosis of recurrent (local or metastatic) disease. If only other cytotoxics were given, they must be stopped at least 4 weeks before randomization. Any hormonal therapy must be stopped at the time of the ICF signature.
* Measurable disease (at least one measurable target lesion assessed by CIR; bone-only or central nervous system [CNS]-only metastases are not allowed).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* LVEF within institutional range of normal at baseline (within 42 days before randomization) as determined by either echocardiography (ECHO) or multigated acquisition (MUGA) scan.
* Adequate hematologic, hepatic and renal function as indicated by the following laboratory values:
* Absolute neutrophil count (ANC) ≥1,500/μL without granulocyte-colony stimulating factor (G-CSF) or other medical support
* Platelets ≥100,000/μL
* Hemoglobin ≥9 g/dL without transfusion or other medical support within 14 days
* Serum creatinine ≤1.5 x upper limit of normal (ULN) and creatinine clearance rate ≥50 mL/min, calculated according to Cockroft-Gault formula
* Serum total bilirubin ≤1.5 x ULN (unless the patient has documented ·Gilbert's syndrome) without any medical support within 14 days
* Serum aspartate aminotransferase/glutamicoxaloacetic transaminase (AST/SGOT) or serum alanine aminotransferase/glutamate-pyruvate transaminase (ALT/SGPT) ≤2.5 x ULN (≤5 x ULN in the case of liver metastases) provided alkaline phosphatase (ALK) is ≤2.5 x ULN. In the case of bone metastasis, serum ALK can be >2.5 x ULN if AST and ALT are ≤1.5 x ULN without any medical support within 14 days
* International normalized ratio (INR), and activated partial prothrombin time (aPTT) or partial prothrombin time (PTT) ≤1.5 x ULN.
* Estimated life expectancy ≥3 months.
* Female patients are eligible to enter and participate in the study if they are of: Non-childbearing potential. Childbearing potential, have a negative serum pregnancy test at Screening, are not breast feeding, and use highly-effective or acceptable contraceptive measures before study entry and throughout the study until 7 months after the last investigational/comparator product administration. Highly-effective or acceptable contraceptive measures.
* Male patients with partners of childbearing potential are eligible to enter and participate in the study if they, and their female partners, are willing to use highly-effective or acceptable contraceptive measures before study entry and throughout the study until 7 months after the last investigational/comparator product administration.

Exclusion Criteria

* Previously- or currently-treated (systemic chemotherapy, biological, or targeted agent, or any other anticancer agent) metastatic breast cancer with the exception of hormonal therapy.
* Known brain metastasis or other CNS metastasis that is either symptomatic or untreated. Central nervous system metastases that have been treated by complete resection and/or radiotherapy demonstrating stability or improvement are not an exclusion criterion provided they are stable as shown by computed tomography (CT) scan for at least 4 weeks before Screening without evidence of cerebral edema and no requirements for corticosteroids or anticonvulsants.
* Participation in another clinical study within 4 weeks before enrollment (3 months for studies involving monoclonal therapy) or the intention of participating in another clinical study during any part of the study period.
* History of other malignancy within the last 5 years, except for carcinoma in-situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin that has been previously treated with curative intent.
* Known history of human immunodeficiency virus (HIV). Clinically significant active infection requiring therapy; positive tests for hepatitis B; or hepatitis C.
* Underlying medical conditions or current severe, uncontrolled systemic disease that, in the Investigator's opinion, will make the administration of study drug hazardous. A major surgical procedure within 4 weeks prior to enrollment or anticipation of the need for major surgery during the course of study.
* Current uncontrolled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg) or unstable angina.
* History of chronic heart failure based on any New York Heart Association (NYHA) criteria, or left ventricular hypertrophy. Current serious cardiac arrhythmia requiring treatment or clinically significant conduction defects as seen on electrocardiogram (ECG). History of myocardial infarction within 6 months of randomization. History of LVEF decline to below 50% during or after previous trastuzumab neo-adjuvant or adjuvant therapy. Significant cardiac murmurs either on examination or ECHO.
* History of prior exposure to doxorubicin >360 mg/m² (or equivalent). Use of oral, injected or implanted hormonal methods of contraception. Chronic daily use of corticoids (equivalent to >10 mg/day methylprednisolone) by oral intake (inhalation is permitted).
* Known hypersensitivity to any of the study drugs.
* Residual non-hematologic toxicity ≥ Grade 2 from prior therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (88):
- China (60):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangzhou University of TMC, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-sen University, Cancer Center, Guanzhou, Guangdong
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Liuzhou General Hospital, Liuchow, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Hebei Cangzhou Central Hospital, Cangzhou, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The 2nd Xiangya Hospital of Central South University, Changsha, Hu'nan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Wuxi 4th People's Hospital, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - General Hospital of the Northern Theater of the Chinese People's Liberation Army, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Qinghai University, Xining, Qinghai
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Jinan Central Hospital, Jinan, Shangdong
  - Yantai Yuhuangding Hospital, Yantai, Shangdong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shannxi Provincial Tumor Hospital, Xi'an, Shangxi
  - The 2nd Hospital of Xi'An Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Nanchong Central Hospital, Nanchong, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing, Tianjing
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Chinese PLA General Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
- Philippines (5):
  - Metro Davao Medical and Research Center, Inc., Davao City, Davao Region
  - Cardinal Santos Medical Center, San Juan City, La Union
  - Manila Doctors Hospital, Manila, National Capital Region
  - The Medical City, Pasig, National Capital Region
  - Cebu Doctors University Hospital, Cebu City
- Ukraine (23):
  - CI Kryvyi Rih Oncological Dispensary of DRC, Kryvyi Rih, Dnepropetrovsk
  - CNE"City Clin Hosp#4"of Dnipro City Council Dept of Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipro, Dnipropetrovsk Oblast
  - CI Carpathian Clinical Oncological Center, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - CNE CCCH of Uzh CC Oncological Center, Ther Dept, SHEI UNU, Uzhhorod, Outer Carpathian
  - Transcarpathian Regional Clinical Oncological Dispensary, Uzhhorod, Outer Carpathian
  - Communal Enterprise Volyn Regional Medical Center of Oncology of Volyn Regional Council, Lutsk, Warren
  - CTPI Chernihiv Regional Oncological Dispensary, Chernihiv
  - CI Chernivtsi RC Oncological Dispensary, Chernivtsi
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv
  - CI of Kherson Reg Council Kherson Regional Oncologic Dispensary, Kherson
  - Khmelnytskyi Regional Oncological Dispensary, Khmelnytskyi
  - Treatment-Diagnostic Center of Private Enterprise of PPC Atsynus, Kropyvnytskyi
  - National Institute of Cancer, Kyiv
  - CNE Kyiv City Clin Oncological Center of Ex Body of Kyiv CC(KCSA), Kyiv
  - Kyiv Сity Clinical Oncological Center, Kyiv
  - CI of LRC Lviv Oncological Regional Treatment and Diagnostic Center, Lviv
  - CI Odesa Regional Clinical Hospital, Odesa
  - Odesa Regional Oncologic Dispensary, Odesa
  - Poltava Reg Cl Onc Dispensary of PRC Chemotherapy Dept HSEI of Ukr UMSA, Poltava
  - RCI Sumy Regional Clinical Oncological Dispensary Dept of of Chemotherapy Sumy SU, Sumy
  - Podilskyi Regional Oncological Center, Vinnytsia
  - CI Zaporizhzhia RC Onc Dispensary of ZRC Dept of Breast Pathology SI Zaporizhzhia MA of PGE of MoHU, Zaporizhzhia
  - CI Zaporizhzhia Regional Clinical Oncological Dispensary of ZRC, Zaporizhzhia

REFERENCES:
- [Derived] Xu B, Zhang Q, Sun T, Li W, Teng Y, Hu X, Bondarenko I, Adamchuk H, Zhang L, Trukhin D, Wang S, Zheng H, Tong Z, Shparyk Y, Yang F, Yu H, Li J, Wang Q, Zhu J; HLX02-BC01 Investigators. Updated efficacy and safety of HLX02 versus reference trastuzumab in metastatic HER2-positive breast cancer: A randomized phase III equivalence trial. Breast. 2025 Apr;80:104413. doi: 10.1016/j.breast.2025.104413. Epub 2025 Feb 4. PMID 39954568
- [Derived] Xu B, Zhang Q, Sun T, Li W, Teng Y, Hu X, Bondarenko I, Adamchuk H, Zhang L, Trukhin D, Wang S, Zheng H, Tong Z, Shparyk Y, Wang Q; HLX02-BC01 Investigators. Efficacy, Safety, and Immunogenicity of HLX02 Compared with Reference Trastuzumab in Patients with Recurrent or Metastatic HER2-Positive Breast Cancer: A Randomized Phase III Equivalence Trial. BioDrugs. 2021 May;35(3):337-350. doi: 10.1007/s40259-021-00475-w. Epub 2021 Apr 7. PMID 33826080

RESULTS

PARTICIPANT FLOW:
Groups:
- HLX02+Docetaxel: HLX02: 8 mg/kg administered intravenously over 90 minutes as a loading dose on Day 1, Cycle 1 then 6 mg/kg every 3 weeks for subsequent cycles for up to a maximum of 12 months.
  Docetaxel: 75 mg/m2 will be administered on Day 2, Cycle 1.then be given every 3 weeks on Day 1 of each subsequent cycle e for at least 8 cycles (until Week 24) and thereafter at the Investigator's discretion for up to a maximum of 12 months.
- Herceptin®+Docetaxel: Herceptin®: 8 mg/kg administered intravenously over 90 minutes as a loading dose on Day 1, Cycle 1 then 6 mg/kg every 3 weeks for subsequent cycles for up to a maximum of 12 months.
  Docetaxel: 75 mg/m2 will be administered on Day 2, Cycle 1.then be given every 3 weeks on Day 1 of each subsequent cycle for at least 8 cycles (until Week 24) and thereafter at the Investigator's discretion for up to a maximum of 12 months.
Period: Overall Study
Arm/Group | HLX02+Docetaxel | Herceptin®+Docetaxel
Started | 325 | 327
Completed | 155 | 137
Not Completed | 170 | 190

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HLX02+Docetaxel | Herceptin®+Docetaxel | Total
Number analyzed (Participants) | 325 | 327 | 652
Age, Continuous [Median (Full Range); unit: years] | 54 [30 to 80] | 53 [26 to 76] | 54 [26 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 325 | 327 | 652
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 249 | 252 | 501
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 76 | 75 | 151
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 238 | 237 | 475
  Philippines | 11 | 15 | 26
  Ukraine | 76 | 75 | 151
ECOG performance status [Count of Participants; unit: Participants]
  0(Fully active, able to carry on all pre-disease performance without restriction) | 138 | 139 | 277
  1(Restricted in physically strenuous activity but ambulatory and able to carry out light work ) | 186 | 186 | 372
  Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: ORR 24
Description: calculated as the proportion of patients with a best response of complete response (CR) or partial response (PR) from first assessment until Week 24 according to RECIST 1.1 by central imaging review (CIR).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions,Complete Response (CR): Disappearance of all target lesions.Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to<10 mm, Partial Response (PR): At least a 30% decrease in the sum ofdiameters of target lesions, taking as reference thebaseline sum diameters.Overall Response (OR) = CR + PR.
Time Frame: From time of First treatment to week 24
Population: ITT set
Measure: Number; unit: percentage of responders
Arm/Group | HLX02+Docetaxel | Herceptin®+Docetaxel
Number analyzed (Participants) | 325 | 327
percentage of responders | 71.1 | 70.9

2. Secondary Outcome: DoR
Description: The time from first documentation of CR or PR to the first documentation of progression.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1)，At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm or Unequivocal progression of existing non-target lesions (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HLX02+Docetaxel | Herceptin®+Docetaxel
Number analyzed (Participants) | 325 | 327
months | 10.61 [10.22 to 11.66] | 10.25 [8.97 to 11.53]

3. Secondary Outcome: DCR
Description: The percentage of patients who achieve CR, PR, or stable disease (SD) of at least 12 weeks
Time Frame: Up to 2 years
Population: ITT set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HLX02+Docetaxel | Herceptin®+Docetaxel
Number analyzed (Participants) | 325 | 327
percentage of participants | 84.3 [80.4 to 88.3] | 87.2 [83.5 to 90.8]

4. Secondary Outcome: CBR
Description: The proportion of patients who achieve CR, PR, or durable SD (SD ≥24 weeks)
Time Frame: Up to 2 years
Population: ITT set
Measure: Number (95% Confidence Interval); unit: Clinical Benefit Rate(%)
Arm/Group | HLX02+Docetaxel | Herceptin®+Docetaxel
Number analyzed (Participants) | 325 | 327
Clinical Benefit Rate(%) | 80.9 [76.7 to 85.2] | 80.4 [76.1 to 84.7]

5. Secondary Outcome: Median PFS up to 12 Months
Description: Median Progression Survival time assessed at 12 months.The probability of being alive without documented progression up to 12 months after randomization.
Time Frame: From time of first treatment to 12 months
Population: ITT set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HLX02+Docetaxel | Herceptin®+Docetaxel
Number analyzed (Participants) | 325 | 327
months | 11.73 [11.53 to 12.06] | 10.55 [9.49 to 11.73]

6. Secondary Outcome: Overall Survival at 12, 24, and 36 Months
Description: the probability of being alive 12, 24, and 36 months after randomization
Time Frame: From time of first treatment to 36 months
Population: ITT set
Measure: Number; unit: percentage of participants with OS
Arm/Group | HLX02+Docetaxel | Herceptin®+Docetaxel
Number analyzed (Participants) | 325 | 327
percentage of participants with OS
  12 months (%) | 88.9 | 88.4
  24 months (%) | 71.4 | 67.6
  36 months (%) | 57.5 | 54.0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date the informed consent form is signed and no later than 30 (+2) days after the last dose, up to 14 months.All-Cause Mortality was assessed up to 36 months.
Arm/Group | HLX02+Docetaxel | Herceptin®+Docetaxel
All-Cause Mortality (participants affected / at risk) | 128/325 | 142/327
Serious Adverse Events (participants affected / at risk) | 78/325 | 81/327
Other Adverse Events (participants affected / at risk) | 320/325 | 321/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HLX02+Docetaxel (N=325) | Herceptin®+Docetaxel (N=327)
Neutrophil count decreased (Investigations) | 33 (58) | 24 (42)
White blood cell count decreased (Investigations) | 16 (31) | 12 (20)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 8 (9) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infusion site infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1)
Puncture site infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (12) | 12 (13)
Myelosuppression (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HLX02+Docetaxel (N=325) | Herceptin®+Docetaxel (N=327)
White blood cell count decreased (Investigations) | 267 (1498) | 276 (1489)
Neutrophil count decreased (Investigations) | 266 (1470) | 268 (1389)
Aspartate aminotransferase increased (Investigations) | 82 (150) | 74 (128)
Alanine aminotransferase increased (Investigations) | 75 (154) | 69 (111)
Weight increased (Investigations) | 48 (60) | 50 (70)
Gamma-glutamyltransferase increased (Investigations) | 37 (62) | 33 (45)
Platelet count decreased (Investigations) | 31 (62) | 33 (56)
Blood alkaline phosphatase increased (Investigations) | 26 (40) | 19 (26)
Weight decreased (Investigations) | 18 (22) | 16 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 181 (182) | 174 (174)
Rash (Skin and subcutaneous tissue disorders) | 32 (43) | 26 (43)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 17 (17) | 20 (21)
Nail discolouration (Skin and subcutaneous tissue disorders) | 13 (13) | 18 (18)
Anaemia (Blood and lymphatic system disorders) | 166 (455) | 187 (498)
Myelosuppression (Blood and lymphatic system disorders) | 20 (53) | 24 (73)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (18) | 20 (21)
Oedema peripheral (General disorders) | 63 (84) | 54 (69)
Pyrexia (General disorders) | 56 (74) | 49 (74)
Asthenia (General disorders) | 31 (51) | 42 (79)
Fatigue (General disorders) | 29 (53) | 30 (55)
Malaise (Blood and lymphatic system disorders) | 30 (44) | 27 (58)
Peripheral swelling (General disorders) | 23 (30) | 21 (28)
Face oedema (General disorders) | 18 (18) | 13 (14)
Diarrhoea (Gastrointestinal disorders) | 76 (163) | 75 (121)
Nausea (Gastrointestinal disorders) | 49 (87) | 58 (94)
Vomiting (Gastrointestinal disorders) | 32 (40) | 35 (48)
Constipation (Gastrointestinal disorders) | 27 (48) | 24 (31)
Stomatitis (Gastrointestinal disorders) | 18 (30) | 21 (56)
Abdominal pain upper (Gastrointestinal disorders) | 12 (13) | 20 (28)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 40 (67) | 45 (89)
Decreased appetite (Metabolism and nutrition disorders) | 35 (48) | 35 (40)
Hypocalcaemia (Metabolism and nutrition disorders) | 29 (61) | 39 (69)
Hypokalaemia (Metabolism and nutrition disorders) | 26 (43) | 30 (41)
Hyperglycaemia (Metabolism and nutrition disorders) | 29 (48) | 18 (43)
Hyperuricaemia (Metabolism and nutrition disorders) | 16 (23) | 29 (49)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12 (18) | 21 (33)
Urinary tract infection (Infections and infestations) | 53 (78) | 61 (102)
Upper respiratory tract infection (Infections and infestations) | 30 (42) | 35 (52)
Pneumonia (Infections and infestations) | 17 (18) | 24 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (60) | 32 (44)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (25) | 19 (30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (23) | 22 (31)
Headache (Nervous system disorders) | 21 (22) | 14 (23)
Dizziness (Nervous system disorders) | 18 (26) | 12 (14)
Infusion related reaction (Injury, poisoning and procedural complications) | 42 (48) | 32 (36)
Insomnia (Psychiatric disorders) | 23 (35) | 27 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT03084237/Prot_SAP_000.pdf